CLINICAL TRIAL: NCT02901626
Title: A Randomized Trial of Pessary in Singleton Pregnancies With a Short Cervix
Acronym: TOPS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped per the recommendation of the DSMB and NICHD.
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HD36801 - TOPS; UG1HD087230 (NIH); UG1HD027915 (NIH); UG1HD034208 (NIH); UG1HD040500 (NIH); UG1HD040485 (NIH); UG1HD053097 (NIH); UG1HD040544 (NIH); UG1HD040545 (NIH); UG1HD040560 (NIH); UG1HD040512 (NIH); UG1HD087192 (NIH); U24HD036801 (NIH); UG1HD027869 (NIH)
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Short Cervix; Preterm Delivery
Keywords: Short cervix; Preterm delivery; Singletons; Pregnancy; Pessary
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The study is an unblinded randomized controlled trial. Participants will receive usual care (vaginal progesterone if they meet criteria per local standard of care) or an Arabin cervical pessary (plus progesterone if the local usual care is to receive vaginal progesterone for a short cervix).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arabin Cervical Pessary (Experimental): Arabin pessary. Participants will also receive vaginal progesterone to be administered daily, if it is the local standard of care.
  Interventions: Device: Arabin Cervical Pessary
- No Pessary (No Intervention): Participants will also receive vaginal progesterone to be administered daily, if it is the local standard of care.

INTERVENTIONS:
Device: Arabin Cervical Pessary — The Arabin cervical pessary is a soft, flexible silicone pessary and fits high around the cervix with no rigid metal framework or inflexible edges that put increase pressure on the vaginal wall. It is available in a variety of sizes however three sizes will be used in this study:
  Pessary Size upper diameter, lower diameter
  1. Nulliparous 65 mm, 32 mm
  2. Multiparous 70 mm, 32 mm
  3. Alternative 70 mm, 35 mm
  Other Names: Arabin pessary
  Arms: Arabin Cervical Pessary

SUMMARY:
The purpose of the study is to determine whether the Arabin pessary is a useful intervention of preterm birth at less than 37 weeks in women with a singleton gestation and a short cervix.

DETAILED DESCRIPTION:
While cervical length is one of the most powerful predictors of subsequent preterm birth, the best treatment to reduce subsequent preterm birth remains unknown. This study is a randomized trial of women who have a singleton pregnancy and a short cervical length on transvaginal ultrasound as determined by a study-certified sonographer. It is being conducted at 12 clinical centers across the country and the recruitment target is enrollment of 850 pregnant women. Participants will be randomized to 1) Arabin pessary or 2) usual care as per by local hospital protocol. Pessary is a promising low-cost, non-surgical intervention that appears to be well-tolerated. The pessary will be placed by obstetric providers trained in appropriate placement of the Arabin pessary. The primary outcome of the study is delivery or fetal death prior to 37 weeks 0 days gestational age.

In the literature, there are two large trials that have produced conflicting results (M Goya et al, 2012, K Nicolaides et al, 2016). Thus, the results of an adequately powered and appropriately conducted trial from the United States will be important in determining whether pessary is a useful intervention for the prevention of subsequent preterm birth in women with singleton gestation.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation. Twin gestation reduced to singleton either spontaneously or therapeutically, is not eligible unless the reduction occurred before 13 weeks 6 days project gestational age. Higher order multifetal gestations reduced to singletons are not eligible.
* Gestational age at randomization between 16 weeks 0 days and 23 weeks 6 days based on clinical information and evaluation of the earliest ultrasound.
* Cervical length on transvaginal examination of less than or equal to 20 mm by a study certified sonographer. There is no lower cervical length threshold.

Exclusion Criteria:

* Cervical dilation (internal os) 3 cm or greater on digital examination or evidence of prolapsed membranes beyond the external cervical os either at the time of the qualifying cervical ultrasound examination or at a cervical exam immediately before randomization.
* Fetal anomaly or imminent fetal demise. This includes lethal anomalies, or anomalies that may lead to early delivery or increased risk of neonatal death e.g., gastroschisis, spina bifida, serious karyotypic abnormalities. An ultrasound examination from 14 weeks 0 days to 23 weeks 6 days by project Estimated Date of Confinement (EDC) must be performed prior to randomization to evaluate the fetus for anomalies.
* Previous spontaneous preterm birth between 16 weeks 0 days and 36 weeks 6 days. This includes induction for pPROM in a prior pregnancy.
* Planned treatment with intramuscular 17-α hydroxy-progesterone caproate.
* Placenta previa, because of risk of bleeding and high potential for indicated preterm birth. A low lying placenta is acceptable.
* Active vaginal bleeding greater than spotting at the time of randomization, because of potential exacerbation due to pessary placement.
* Symptomatic, untreated vaginal or cervical infection because of potential exacerbation due to pessary placement. Patients may be treated and if subsequently asymptomatic, randomized. However, if it is more than 10 days since the cervical length measurement, a new cervical length measurement must be obtained.
* Active, unhealed herpetic lesion on labia minora, vagina, or cervix due to the potential for significant patient discomfort or increasing genital tract viral spread. Once lesion(s) heal and the patient is asymptomatic, she may be randomized. History of herpes is not an exclusion.
* Rupture of membranes due to likelihood of pregnancy loss and preterm delivery as well as the risk of ascending infection which could be increased with pessary placement.
* More than six contractions per hour reported or documented prior to randomization. It is not necessary to place the patient on a tocodynamometer.
* Known major Mullerian anomaly of the uterus (specifically bicornuate, unicornuate, or uterine septum not resected) due to increased risk of preterm delivery which is unlikely to be affected by progesterone.
* Any fetal/maternal condition which would require invasive in-utero assessment or treatment, for example significant red cell antigen sensitization or neonatal alloimmune thrombocytopenia.
* Major maternal medical illness associated with increased risk for adverse pregnancy outcome or indicated preterm birth (treated hypertension requiring more than one agent, treatment for diabetes prior to pregnancy, chronic renal insufficiency defined by creatinine >1.4 mg/dL, carcinoma of the breast, conditions treated with chronic oral glucocorticoid therapy). Lupus, uncontrolled thyroid disease, and New York Heart Association(NYHA) stage II or greater cardiac disease are also excluded. Patients with seizure disorders, HIV, and other medical conditions not specifically associated with an increased risk of indicated preterm birth are not excluded. Prior cervical cone/LOOP/Loop Electrocautery Excision Procedure (LEEP) is not an exclusion criterion.
* Planned cerclage or cerclage already in place since it would preclude placement of a pessary.
* Planned indicated delivery prior to 37 weeks.
* Allergy to silicone.
* Participation in another interventional study that influences gestational age at delivery or neonatal morbidity or mortality.
* Participation in this trial in a previous pregnancy. Patients who were screened in a previous pregnancy, but not randomized, may be included.
* Prenatal care or delivery planned elsewhere unless the study visits can be made as scheduled and complete outcome information can be obtained.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Clifton, Ph.D., Principal Investigator — George Washington University Biostatistics Center; Monica Longo, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Matthew Hoffman, MD, Study Chair — Christiana Care Health Services
Locations (12):
- United States (12):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Womens, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after the completion of the trial and publication of the main analyses per NIH policy. Data will be available through the NICHD Data and Specimen Hub
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Hamilton BE, Martin JA, Osterman MJ, Curtin SC, Matthews TJ. Births: Final Data for 2014. Natl Vital Stat Rep. 2015 Dec;64(12):1-64. PMID 26727629
- [Background] Lawn JE, Kerber K, Enweronu-Laryea C, Cousens S. 3.6 million neonatal deaths--what is progressing and what is not? Semin Perinatol. 2010 Dec;34(6):371-86. doi: 10.1053/j.semperi.2010.09.011. PMID 21094412
- [Background] American College of Obstetricians and Gynecologists; Committee on Practice Bulletins-Obstetrics. ACOG practice bulletin no. 127: Management of preterm labor. Obstet Gynecol. 2012 Jun;119(6):1308-17. doi: 10.1097/AOG.0b013e31825af2f0. PMID 22617615
- [Background] Meis PJ, Klebanoff M, Thom E, Dombrowski MP, Sibai B, Moawad AH, Spong CY, Hauth JC, Miodovnik M, Varner MW, Leveno KJ, Caritis SN, Iams JD, Wapner RJ, Conway D, O'Sullivan MJ, Carpenter M, Mercer B, Ramin SM, Thorp JM, Peaceman AM, Gabbe S; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Prevention of recurrent preterm delivery by 17 alpha-hydroxyprogesterone caproate. N Engl J Med. 2003 Jun 12;348(24):2379-85. doi: 10.1056/NEJMoa035140. PMID 12802023
- [Background] da Fonseca EB, Bittar RE, Carvalho MH, Zugaib M. Prophylactic administration of progesterone by vaginal suppository to reduce the incidence of spontaneous preterm birth in women at increased risk: a randomized placebo-controlled double-blind study. Am J Obstet Gynecol. 2003 Feb;188(2):419-24. doi: 10.1067/mob.2003.41. PMID 12592250
- [Background] Petrini JR, Callaghan WM, Klebanoff M, Green NS, Lackritz EM, Howse JL, Schwarz RH, Damus K. Estimated effect of 17 alpha-hydroxyprogesterone caproate on preterm birth in the United States. Obstet Gynecol. 2005 Feb;105(2):267-72. doi: 10.1097/01.AOG.0000150560.24297.4f. PMID 15684150
- [Background] Andersen HF, Nugent CE, Wanty SD, Hayashi RH. Prediction of risk for preterm delivery by ultrasonographic measurement of cervical length. Am J Obstet Gynecol. 1990 Sep;163(3):859-67. doi: 10.1016/0002-9378(90)91084-p. PMID 2206073
- [Background] Iams JD, Goldenberg RL, Meis PJ, Mercer BM, Moawad A, Das A, Thom E, McNellis D, Copper RL, Johnson F, Roberts JM. The length of the cervix and the risk of spontaneous premature delivery. National Institute of Child Health and Human Development Maternal Fetal Medicine Unit Network. N Engl J Med. 1996 Feb 29;334(9):567-72. doi: 10.1056/NEJM199602293340904. PMID 8569824
- [Background] Heath VC, Southall TR, Souka AP, Elisseou A, Nicolaides KH. Cervical length at 23 weeks of gestation: prediction of spontaneous preterm delivery. Ultrasound Obstet Gynecol. 1998 Nov;12(5):312-7. doi: 10.1046/j.1469-0705.1998.12050312.x. PMID 9819868
- [Background] Fonseca EB, Celik E, Parra M, Singh M, Nicolaides KH; Fetal Medicine Foundation Second Trimester Screening Group. Progesterone and the risk of preterm birth among women with a short cervix. N Engl J Med. 2007 Aug 2;357(5):462-9. doi: 10.1056/NEJMoa067815. PMID 17671254
- [Background] O'Brien JM, Adair CD, Lewis DF, Hall DR, Defranco EA, Fusey S, Soma-Pillay P, Porter K, How H, Schackis R, Eller D, Trivedi Y, Vanburen G, Khandelwal M, Trofatter K, Vidyadhari D, Vijayaraghavan J, Weeks J, Dattel B, Newton E, Chazotte C, Valenzuela G, Calda P, Bsharat M, Creasy GW. Progesterone vaginal gel for the reduction of recurrent preterm birth: primary results from a randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2007 Oct;30(5):687-96. doi: 10.1002/uog.5158. PMID 17899572
- [Background] Hassan SS, Romero R, Vidyadhari D, Fusey S, Baxter JK, Khandelwal M, Vijayaraghavan J, Trivedi Y, Soma-Pillay P, Sambarey P, Dayal A, Potapov V, O'Brien J, Astakhov V, Yuzko O, Kinzler W, Dattel B, Sehdev H, Mazheika L, Manchulenko D, Gervasi MT, Sullivan L, Conde-Agudelo A, Phillips JA, Creasy GW; PREGNANT Trial. Vaginal progesterone reduces the rate of preterm birth in women with a sonographic short cervix: a multicenter, randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2011 Jul;38(1):18-31. doi: 10.1002/uog.9017. Epub 2011 Jun 15. PMID 21472815
- [Background] Romero R, Nicolaides K, Conde-Agudelo A, Tabor A, O'Brien JM, Cetingoz E, Da Fonseca E, Creasy GW, Klein K, Rode L, Soma-Pillay P, Fusey S, Cam C, Alfirevic Z, Hassan SS. Vaginal progesterone in women with an asymptomatic sonographic short cervix in the midtrimester decreases preterm delivery and neonatal morbidity: a systematic review and metaanalysis of individual patient data. Am J Obstet Gynecol. 2012 Feb;206(2):124.e1-19. doi: 10.1016/j.ajog.2011.12.003. Epub 2011 Dec 11. PMID 22284156
- [Background] Grobman WA, Thom EA, Spong CY, Iams JD, Saade GR, Mercer BM, Tita AT, Rouse DJ, Sorokin Y, Wapner RJ, Leveno KJ, Blackwell S, Esplin MS, Tolosa JE, Thorp JM Jr, Caritis SN, Van Dorsten JP; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units (MFMU) Network. 17 alpha-hydroxyprogesterone caproate to prevent prematurity in nulliparas with cervical length less than 30 mm. Am J Obstet Gynecol. 2012 Nov;207(5):390.e1-8. doi: 10.1016/j.ajog.2012.09.013. Epub 2012 Sep 17. PMID 23010094
- [Background] Norman JE, Marlow N, Messow CM, Shennan A, Bennett PR, Thornton S, Robson SC, McConnachie A, Petrou S, Sebire NJ, Lavender T, Whyte S, Norrie J; OPPTIMUM study group. Vaginal progesterone prophylaxis for preterm birth (the OPPTIMUM study): a multicentre, randomised, double-blind trial. Lancet. 2016 May 21;387(10033):2106-2116. doi: 10.1016/S0140-6736(16)00350-0. Epub 2016 Feb 24. PMID 26921136
- [Background] Committee on Practice Bulletins-Obstetrics, The American College of Obstetricians and Gynecologists. Practice bulletin no. 130: prediction and prevention of preterm birth. Obstet Gynecol. 2012 Oct;120(4):964-73. doi: 10.1097/AOG.0b013e3182723b1b. No abstract available. PMID 22996126
- [Background] Society for Maternal-Fetal Medicine Publications Committee, with assistance of Vincenzo Berghella. Progesterone and preterm birth prevention: translating clinical trials data into clinical practice. Am J Obstet Gynecol. 2012 May;206(5):376-86. doi: 10.1016/j.ajog.2012.03.010. PMID 22542113
- [Background] Cahill AG, Odibo AO, Caughey AB, Stamilio DM, Hassan SS, Macones GA, Romero R. Universal cervical length screening and treatment with vaginal progesterone to prevent preterm birth: a decision and economic analysis. Am J Obstet Gynecol. 2010 Jun;202(6):548.e1-8. doi: 10.1016/j.ajog.2009.12.005. Epub 2010 Jan 15. PMID 20079888
- [Background] Werner EF, Han CS, Pettker CM, Buhimschi CS, Copel JA, Funai EF, Thung SF. Universal cervical-length screening to prevent preterm birth: a cost-effectiveness analysis. Ultrasound Obstet Gynecol. 2011 Jul;38(1):32-7. doi: 10.1002/uog.8911. Epub 2011 May 24. PMID 21157771
- [Background] Berghella V, Odibo AO, To MS, Rust OA, Althuisius SM. Cerclage for short cervix on ultrasonography: meta-analysis of trials using individual patient-level data. Obstet Gynecol. 2005 Jul;106(1):181-9. doi: 10.1097/01.AOG.0000168435.17200.53. PMID 15994635
- [Background] Owen J, Hankins G, Iams JD, Berghella V, Sheffield JS, Perez-Delboy A, Egerman RS, Wing DA, Tomlinson M, Silver R, Ramin SM, Guzman ER, Gordon M, How HY, Knudtson EJ, Szychowski JM, Cliver S, Hauth JC. Multicenter randomized trial of cerclage for preterm birth prevention in high-risk women with shortened midtrimester cervical length. Am J Obstet Gynecol. 2009 Oct;201(4):375.e1-8. doi: 10.1016/j.ajog.2009.08.015. PMID 19788970
- [Background] Arabin B, Halbesma JR, Vork F, Hubener M, van Eyck J. Is treatment with vaginal pessaries an option in patients with a sonographically detected short cervix? J Perinat Med. 2003;31(2):122-33. doi: 10.1515/JPM.2003.017. PMID 12747228
- [Background] Goya M, Pratcorona L, Merced C, Rodo C, Valle L, Romero A, Juan M, Rodriguez A, Munoz B, Santacruz B, Bello-Munoz JC, Llurba E, Higueras T, Cabero L, Carreras E; Pesario Cervical para Evitar Prematuridad (PECEP) Trial Group. Cervical pessary in pregnant women with a short cervix (PECEP): an open-label randomised controlled trial. Lancet. 2012 May 12;379(9828):1800-6. doi: 10.1016/S0140-6736(12)60030-0. Epub 2012 Apr 3. PMID 22475493
- [Background] Nicolaides KH, Syngelaki A, Poon LC, Picciarelli G, Tul N, Zamprakou A, Skyfta E, Parra-Cordero M, Palma-Dias R, Rodriguez Calvo J. A Randomized Trial of a Cervical Pessary to Prevent Preterm Singleton Birth. N Engl J Med. 2016 Mar 17;374(11):1044-52. doi: 10.1056/NEJMoa1511014. PMID 26981934
- [Background] Hui SY, Chor CM, Lau TK, Lao TT, Leung TY. Cerclage pessary for preventing preterm birth in women with a singleton pregnancy and a short cervix at 20 to 24 weeks: a randomized controlled trial. Am J Perinatol. 2013 Apr;30(4):283-8. doi: 10.1055/s-0032-1322550. Epub 2012 Aug 8. PMID 22875662
- [Background] Gyamfi-Bannerman C, Ananth CV. Trends in spontaneous and indicated preterm delivery among singleton gestations in the United States, 2005-2012. Obstet Gynecol. 2014 Dec;124(6):1069-1074. doi: 10.1097/AOG.0000000000000546. PMID 25415156
- [Background] Committee opinion no 611: method for estimating due date. Obstet Gynecol. 2014 Oct;124(4):863-866. doi: 10.1097/01.AOG.0000454932.15177.be. PMID 25244460
- [Background] Conde-Agudelo A, Romero R, Nicolaides K, Chaiworapongsa T, O'Brien JM, Cetingoz E, da Fonseca E, Creasy G, Soma-Pillay P, Fusey S, Cam C, Alfirevic Z, Hassan SS. Vaginal progesterone vs. cervical cerclage for the prevention of preterm birth in women with a sonographic short cervix, previous preterm birth, and singleton gestation: a systematic review and indirect comparison metaanalysis. Am J Obstet Gynecol. 2013 Jan;208(1):42.e1-42.e18. doi: 10.1016/j.ajog.2012.10.877. Epub 2012 Nov 15. PMID 23157855
- [Background] Lan KK, Wittes J. The B-value: a tool for monitoring data. Biometrics. 1988 Jun;44(2):579-85. PMID 3390511
- [Background] Stallones RA. The use and abuse of subgroup analysis in epidemiological research. Prev Med. 1987 Mar;16(2):183-94. doi: 10.1016/0091-7435(87)90082-x. PMID 3295858
- [Background] Yusuf S, Wittes J, Probstfield J, Tyroler HA. Analysis and interpretation of treatment effects in subgroups of patients in randomized clinical trials. JAMA. 1991 Jul 3;266(1):93-8. PMID 2046134
- [Background] Facco FL, Simhan HN. Short ultrasonographic cervical length in women with low-risk obstetric history. Obstet Gynecol. 2013 Oct;122(4):858-862. doi: 10.1097/AOG.0b013e3182a2dccd. PMID 24084545
- [Derived] Hoffman MK, Clifton RG, Biggio JR, Saade GR, Ugwu LG, Longo M, Bousleiman SZ, Clark K, Grobman WA, Frey HA, Chauhan SP, Dugoff L, Manuck TA, Chien EK, Rouse DJ, Simhan HN, Esplin MS, Macones GA; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units (MFMU) Network. Cervical Pessary for Prevention of Preterm Birth in Individuals With a Short Cervix: The TOPS Randomized Clinical Trial. JAMA. 2023 Jul 25;330(4):340-348. doi: 10.1001/jama.2023.10812. PMID 37490086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2017 through November 5, 2021 we conducted a multicenter randomized trial comparing the Arabin pessary versus usual care at 12 clinical centers. Individuals with asymptomatic singleton pregnancies who had a transvaginal cervical length <20mm between 16 weeks 0 days and 23 weeks 6 days were identified per the local protocol for assessment of cervical length. People meeting eligibility requirements and accepting trial participation were randomized to either pessary or usual care.
Groups:
- Arabin Cervical Pessary: Arabin pessary. Participants will also receive vaginal progesterone to be administered daily, if it is the local standard of care.
  Pessary: The Arabin cervical pessary is a soft, flexible silicone pessary and fits high around the cervix with no rigid metal framework or inflexible edges that put increase pressure on the vaginal wall. It is available in a variety of sizes however three sizes will be used in this study:
  Pessary Size upper diameter, lower diameter
  1. Nulliparous 65 mm, 32 mm
  2. Multiparous 70 mm, 32 mm
  3. Alternative 70 mm, 35 mm
Period: Overall Study
Arm/Group | Arabin Cervical Pessary | No Pessary
Started | 280 | 264
Completed | 279 | 263
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cervical Arabin Pessary: Arabin pessary. Participants will also receive vaginal progesterone to be administered daily, if it is the local standard of care.
  Pessary: The Arabin cervical pessary is a soft, flexible silicone pessary and fits high around the cervix with no rigid metal framework or inflexible edges that put increase pressure on the vaginal wall. It is available in a variety of sizes however three sizes will be used in this study:
  Pessary Size upper diameter, lower diameter
  1. Nulliparous 65 mm, 32 mm
  2. Multiparous 70 mm, 32 mm
  3. Alternative 70 mm, 35 mm
- Total: Total of all reporting groups
Arm/Group | Cervical Arabin Pessary | No Pessary | Total
Number analyzed (Participants) | 280 | 264 | 544
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (6.0) | 29.1 (5.9) | 29.5 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280 | 264 | 544
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Black | 132 | 127 | 259
  Non-Hispanic White | 61 | 53 | 114
  Hispanic | 62 | 56 | 118
  Asian | 12 | 16 | 28
  Native Hawaiian/Pacific Islander | 0 | 1 | 1
  American Indian | 1 | 0 | 1
  Other/not reported/unknown | 12 | 11 | 23
Gestational age at enrollment (weeks) [Median (Inter-Quartile Range); unit: weeks] | 21.7 [20.6 to 22.9] | 21.9 [20.7 to 23.2] | 21.7 [20.7 to 23.0]
Cervical length at screening (mm) [Mean (Standard Deviation); unit: mm] | 12.7 (5.2) | 12.7 (5.3) | 12.7 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Preterm Delivery or Fetal Death at Less Than 37 Weeks.
Description: Participants who either delivered or experienced a fetal death prior to 37 weeks gestation.
Time Frame: Before 37 weeks 0 days gestation, a period of up to 21 weeks from enrollment.
Population: 1 participant in each group was lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
Participants | 127 | 120
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.83 to 1.20]

2. Secondary Outcome: Interval From Randomization to Delivery or Fetal Death
Description: The median interval between randomization to delivery or death of the fetus.
Time Frame: from randomization to delivery or fetal death (up to a length of 189 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
days | 105 [42 to 120] | 103 [56 to 118]
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Median Difference (Net) = 2, 95% CI 2-sided [-4 to 8]

3. Secondary Outcome: Gestational Age at Delivery
Description: Median gestational age (in weeks) at the time of delivery
Time Frame: From randomization to delivery (up to a length of 189 days)
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Arabin Cervical Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
weeks | 37.3 [27.4 to 39.1] | 37.4 [29.6 to 39.1]
Statistical Analysis 1: Comparison: Arabin Cervical Pessary vs No Pessary; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.06 to 0.80]

4. Secondary Outcome: Number of Participants With Preterm Delivery or Fetal Death at Less Than 28 Weeks Gestation
Description: The number of participants who either delivered or experienced a fetal death prior to 28 weeks gestation.
Time Frame: from randomization to less than 28 weeks gestation (a period of less than 91 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
Participants | 72 | 54
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.26, 95% CI 2-sided [0.92 to 1.71]

5. Secondary Outcome: Number of Participants With Preterm Delivery or Fetal Death at Less Than 32 Weeks Gestation
Description: The number of participants who either delivered or experienced a fetal death prior to 32 weeks gestation.
Time Frame: from randomization to less than 32 weeks gestation (a period of less than 119 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
Participants | 93 | 73
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.20, 95% CI 2-sided [0.93 to 1.55]

6. Secondary Outcome: Number of Participants With Preterm Delivery or Fetal Death at Less Than 35 Weeks Gestation
Description: The number of participants who either delivered or experienced a fetal death prior to 35 weeks gestation.
Time Frame: from randomization to less than 35 weeks gestation (a period of less than 140 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
Participants | 111 | 90
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.93 to 1.45]

7. Secondary Outcome: Number of Participants With Preterm Premature Rupture of Membranes
Description: Participants were categorized as yes if the amniotic membranes ruptured prior to labor onset and before 37 weeks gestation.
Time Frame: Before 37 weeks 0 days gestation, a period of up to 21 weeks from enrollment
Population: Data is missing for 2 participants in the pessary group and 5 participants in the no pessary group.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 277 | 258
Participants | 64 | 46
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.30, 95% CI 2-sided [0.92 to 1.82]

8. Secondary Outcome: Number of Participants With Spontaneous Preterm Delivery.
Description: The number of participants who experienced spontaneous onset of labor and had an unassisted vaginal delivery prior to 37 weeks gestation. Induction for delivery was not performed and operative techniques such as forceps or vacuum were not used.
Time Frame: From randomization to delivery (up to a length of 189 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
Participants | 109 | 106
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.79 to 1.19]

9. Secondary Outcome: Number of Participants With Indicated Preterm Delivery
Description: The number of participants who underwent labor induction or had an assisted vaginal delivery with forceps or vacuum or cesarean delivery prior to 37 weeks gestation.
Time Frame: from randomization to delivery (up to a length of 189 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
Participants | 18 | 14
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.61 to 2.39]

10. Secondary Outcome: Number of Participants With Cesarean Delivery
Description: The number of participants who underwent a surgical procedure for delivery (cesarean) at any gestational age.
Time Frame: From randomization to delivery (up to a length of 189 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
Participants | 86 | 80
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.79 to 1.31]

11. Secondary Outcome: Number of Participants With Chorioamnionitis
Description: The number of participants who had a clinical diagnosis of chorioamnionitis and a body temperature of at least 100.0° F (38° C) and no other defined infection.
Time Frame: From randomization to delivery (up to a length of 189 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
Participants | 18 | 16
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.55 to 2.04]

12. Secondary Outcome: Median Length of Maternal Antepartum Hospital Stay Before Delivery
Description: Median number of days from maternal hospital admission for delivery and the date of delivery.
Time Frame: from date of admission for delivery up to delivery date (up to 5 days)
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Pessary: Arabin pessary. Participants will also receive vaginal progesterone to be administered daily, if it is the local standard of care.
  Pessary: The Arabin cervical pessary is a soft, flexible silicone pessary and fits high around the cervix with no rigid metal framework or inflexible edges that put increase pressure on the vaginal wall. It is available in a variety of sizes however three sizes will be used in this study:
  Pessary Size upper diameter, lower diameter
  1. Nulliparous 65 mm, 32 mm
  2. Multiparous 70 mm, 32 mm
  3. Alternative 70 mm, 35 mm
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 279 | 263
days | 1 [0 to 1] | 1 [0 to 1]
Statistical Analysis 1: Comparison: Pessary vs No Pessary; Test type: Superiority; Median Difference (Net) = 0, 95% CI 2-sided [0 to 0]

13. Secondary Outcome: Number of Participants With Vaginal Infection
Description: The number of participants with a clinical diagnosis of a vaginal infection. Includes participants with at least one study visit.
Time Frame: From randomization to delivery (up to a length of 189 days)
Population: Data missing for 53 participants in the pessary group and 43 participants in the no pessary group.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 226 | 220
Participants | 57 | 41
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.36, 95% CI 2-sided [0.95 to 1.94]

14. Secondary Outcome: The Number of Participants Who Had a Vaginal Infection and Received Antibiotic Treatment, Among All Persons Enrolled With at Least One Study Visit
Description: The number of participants who received antibiotics or antifungal medication for a vaginal infection (out of the total sample for which data is available)
Time Frame: From randomization to delivery (up to a length of 189 days)
Population: Data missing for 53 participants in the pessary group and 43 participants in the no pessary group.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 226 | 220
Participants | 55 | 37
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.45, 95% CI 2-sided [1.00 to 2.11]

15. Secondary Outcome: Number of Participants Treated for Preterm Labor Including Placement of Cerclage
Description: The number of participants who received any one of the following treatments for preterm labor: tocolysis, cerclage, bedrest, antenatal corticosteroids for fetal lung maturity, or magnesium sulfate for neuroprotection.
Time Frame: From randomization to delivery (up to a length of 189 days)
Population: Data missing for 21 participants in the pessary group and 13 participants in the no pessary group.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 258 | 250
Participants | 150 | 143
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.88 to 1.18]

16. Secondary Outcome: Median Duration of Neonatal Ventilator or Continuous Positive Airway Pressure Use
Description: Median number of days a neonate or infant was on a ventilator or received continuous positive airway pressure.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 97 | 104
days | 6 [0 to 43] | 5 [0 to 41]
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Median Difference (Net) = 0, 95% CI 2-sided [-12 to 12]

17. Secondary Outcome: Number of Neonates Requiring Ventilator or Continuous Positive Airway Pressure Use
Description: The number of neonates or infants who required ventilator support or received continuous positive airway pressure.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9). 2 neonates missing date in the pessary group
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 254
Participants | 75 | 82
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.69 to 1.17]

18. Secondary Outcome: Median Duration (in Days) of Neonatal Supplemental Oxygen Use
Description: Median number of days a neonate received supplemental oxygen after admission to the NICU or intermediate nursery. Supplemental oxygen is defined as FiO2 > 0.21.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 95 | 105
days | 7 [0 to 41] | 6 [0 to 51]
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Median Difference (Net) = 1, 95% CI 2-sided [-12 to 14]

19. Secondary Outcome: Number of Neonates With Seizures Requiring Treatment
Description: The number of neonates with a clinical diagnosis of seizures who received anti-seizure medication.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 254
Participants | 1 | 1
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.06 to 15.7]

20. Secondary Outcome: Number of Neonates Small for Gestational Age < 5th Percentile
Description: The number of neonates whose birthweight compared with gestational age at delivery was less than the 5th percentile, as assessed by sex and race, using United States birth certificate data.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 258 | 253
Participants | 5 | 6
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.25 to 2.65]

21. Secondary Outcome: Number of Neonates With Intraventricular Hemorrhage (IVH) Grades III or IV
Description: IVH grades III or IV are as determined by cranial ultrasounds performed as part of routine clinical care and classified based on the Papile classification system
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9). there are 3 neonates with missing data in the pessary group.
Measure: Count of Participants; unit: Participants
Groups:
- Cervical Arabin Pessary: Arabin pessary. Participants will also receive vaginal progesterone to be administered daily, if it is the local standard of .
  Pessary: The Arabin cervical pessary is a soft, flexible silicone pessary and fits high around the cervix with no rigid metal framework or inflexible edges that put increase pressure on the vaginal wall. It is available in a variety of sizes however three sizes will be used in this study:
  Pessary Size upper diameter, lower diameter
  1. Nulliparous 65 mm, 32 mm
  2. Multiparous 70 mm, 32 mm
  3. Alternative 70 mm, 35 mm
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 258 | 254
Participants | 4 | 7
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.56, 95% CI 2-sided [0.17 to 1.90]

22. Secondary Outcome: Number of Neonates With Retinopathy of Prematurity (ROP)
Description: The number of neonates with a clinical diagnosis of retinopathy of prematurity where an ophthalmologic examination of the retina was performed.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9). 2 neonates in the pessary group are missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 254
Participants | 27 | 23
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.15, 95% CI 2-sided [0.68 to 1.96]

23. Secondary Outcome: Number of Neonates Experiencing Respiratory Distress Syndrome (RDS)
Description: The number of neonates with a diagnosis of respiratory distress syndrome defined as the presence of clinical signs of respiratory distress (tachypnea, retractions, flaring, grunting, or cyanosis), with oxygen requirement and a chest x-ray that show hypoaeration and reticulogranular infiltrates.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 254
Participants | 67 | 69
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.71 to 1.27]

24. Secondary Outcome: Number of Neonates With Bronchopulmonary Dysplasia (BPD)
Description: The number of neonates with a clinical diagnosis of bronchopulmonary dysplasia defined as oxygen requirement at 28 days of life if delivered at or after 32 weeks gestation, or at 36 weeks project gestational age if delivered before 32 weeks gestation.
Time Frame: Delivery through 28 days of life if delivered at or after 32 weeks. Delivery through 36 weeks gestation if delivered before 32 weeks.
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 260 | 254
Participants | 14 | 19
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.72, 95% CI 2-sided [0.37 to 1.41]

25. Secondary Outcome: Number of Neonates With Necrotizing Enterocolitis (NEC) Stage 2 or 3
Description: The number of neonates diagnosed with NEC, defined as modified Bell Stage 2 or 3 where stage 2 represents clinical signs and symptoms with pneumatosis intestinalis on radiographs and stage 3 is defined as advanced clinical signs and symptoms, pneumatosis, impending or proven intestinal perforation.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 254
Participants | 7 | 6
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.39 to 3.37]

26. Secondary Outcome: Number of Neonates With Hyperbilirubinemia
Description: The number of neonates diagnosed with hyperbilirubinemia, defined as peak total bilirubin of at least 15 mg% or the use of phototherapy
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9). 2 neonates missing data in the pessary group. 1 neonate missing data in the no pessary group.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 253
Participants | 84 | 82
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.78 to 1.29]

27. Secondary Outcome: Neonatal Infectious Morbidity Including Sepsis, Suspected Sepsis and Pneumonia
Description: The number of neonates diagnosed with any one of the following:
  * Sepsis (within 72 hours and > 72 hours after birth) defined as a clinically ill infant in whom systemic infection is suspected with a positive blood, CSF, or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an unequivocal radiograph confirming infection.
  * Suspected sepsis. The diagnosis of suspected sepsis will include infants with suspicious clinical findings of infection, but no positive cultures or radiographs.
  * Pneumonia. The diagnosis of pneumonia will be confirmed by radiograph or positive blood culture.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9). 2 neonates missing data in the pessary group
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 254
Participants | 53 | 65
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.58 to 1.10]

28. Secondary Outcome: Number of Neonates With Early Onset Sepsis
Description: The number of neonates with a clinical diagnosis of sepsis within 72 hours of life, defined as a clinically ill infant in whom systemic infection is suspected with a positive blood, cerebrospinal fluid, or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an unequivocal radiograph confirming infection.
Time Frame: within 72 hours of birth
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 254
Participants | 5 | 2
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 2.45, 95% CI 2-sided [0.48 to 12.57]

29. Secondary Outcome: Number of Neonates With Late Onset Sepsis
Description: The number of neonates with a clinical diagnosis of sepsis at or after 72 hours of life, defined as the presence of a clinically ill infant in whom systemic infection is suspected with a positive blood, cerebrospinal fluid, or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an unequivocal radiograph confirming infection.
Time Frame: 72 hours of birth or later (up to hospital discharge - a maximum of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 254
Participants | 8 | 12
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.65, 95% CI 2-sided [0.27 to 1.58]

30. Secondary Outcome: Number of Neonates With Suspected Sepsis
Description: The number of neonates with suspicious clinical findings of infection, but no positive cultures or radiographs.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 254
Participants | 38 | 51
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.47 to 0.97]

31. Secondary Outcome: Number of Neonates With Pneumonia
Description: The number of neonates with a clinical diagnosis of pneumonia within 72 hours of birth and confirmed by either an x-ray demonstrating consolidation with air bronchograms, or a positive blood culture performed at the time of clinical diagnosis.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 259 | 254
Participants | 2 | 4
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 0.49, 95% CI 2-sided [0.09 to 2.66]

32. Secondary Outcome: Number of Neonates With Composite Outcome
Description: The number of neonates diagnosed with any one of fetal or neonatal death or Respiratory Distress Syndrome, Grade 3 or 4 Intraventricular Hemorrhage, Periventricular Leukomalacia, Stage 2 or 3 Nectrotizing Enterocolitis, Bronchopulmonary Dysplasia, Stage III or higher Retinopathy of Prematurity, or early onset sepsis.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9). 1 neonate missing data in the pessary group
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 260 | 254
Participants | 81 | 74
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.81 to 1.37]

33. Secondary Outcome: Median Length of Neonatal Hospital Stay
Description: Median number of days the neonate/infant remained in hospital.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 258 | 253
days | 3 [2 to 20] | 3 [2 to 22]
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Median Difference (Net) = 0, 95% CI 2-sided [0 to 0]

34. Secondary Outcome: Median Number of Days in Neonatal Intensive Care Unit (NICU)
Description: Median number of days the neonate/infant remained in the neonatal intensive care unit or special care nursery.
Time Frame: delivery through hospital discharge (up to a length of 435 days)
Population: among livebirth deliveries (excludes fetal deaths - pessary 18, no pessary 9)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cervical Arabin Pessary | No Pessary
Number analyzed (Participants) | 97 | 104
days | 50 [10 to 99] | 37 [11 to 88]
Statistical Analysis 1: Comparison: Cervical Arabin Pessary vs No Pessary; Test type: Superiority; Median Difference (Net) = 10, 95% CI 2-sided [-16 to 36]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from from delivery (up to 175 days after randomization) through hospital discharge of the neonate (up to a length of 435 days). All cause mortality was assessed from delivery to 28 days after the expected date of delivery, if discharged from hospital on or before 28 days after the expected date of delivery. If discharged from hospital after 28 days after the expected date of delivery, all cause mortality was assessed from delivery to hospital discharge.
Groups:
- Cervical Arabin Pessary: Arabin pessary. Participants will also receive vaginal progesterone to be administered daily, if it is the local standard of care.
Arm/Group | Cervical Arabin Pessary | No Pessary
All-Cause Mortality (participants affected / at risk) | 37/280 | 18/264
Serious Adverse Events (participants affected / at risk) | 13/280 | 17/264
Other Adverse Events (participants affected / at risk) | 248/280 | 200/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervical Arabin Pessary (N=280) | No Pessary (N=264)
Hypertension Management (Vascular disorders) | 0 (0) | 1 (1) — hospitalized for adjustment of BP meds after not taking meds as prescribed
Neonatal ventricular septal defect (Vascular disorders) | 1 (1) | 1 (1)
Neonatal intestinal failure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glucoregulation in the setting of steroid administration (Endocrine disorders) | 0 (0) | 1 (1) — hospitalized for management of gestational diabetes (along with antenatal corticosteroids)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinemia and weight loss (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sars-CoV-2 Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — maternal COVID-19 infection
Hospital-based pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory syncytial virus/ bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal central nervous system malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ambiguous genitalia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypospadias (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Post-partum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Neonatal amputation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Auditory hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic multifocal osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neonatal CN6 Palsy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Disseminated herpes simplex virus (Infections and infestations) | 1 (1) | 0 (0)
Erb-Duchenne Palsy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neonatal hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Trisomy 21 (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Necrotizing enterocolitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervical Arabin Pessary (N=280) | No Pessary (N=264)
Vaginal fluid leakage (Pregnancy, puerperium and perinatal conditions) | 26 (27) | 2 (2)
Lower abdominal/pelvic pain (Pregnancy, puerperium and perinatal conditions) | 79 (118) | 80 (124)
Lower abdominal/pelvic pressure (Pregnancy, puerperium and perinatal conditions) | 103 (190) | 89 (165)
Urinary change in frequency and incontinence (Pregnancy, puerperium and perinatal conditions) | 53 (78) | 37 (53)
Vaginal bleeding (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 15 (15)
Vaginal burning (Pregnancy, puerperium and perinatal conditions) | 21 (27) | 16 (19)
Vaginal discharge (Pregnancy, puerperium and perinatal conditions) | 201 (477) | 160 (321)
Vaginal discomfort/soreness (Pregnancy, puerperium and perinatal conditions) | 101 (175) | 69 (119)
Vaginal itching (Pregnancy, puerperium and perinatal conditions) | 45 (72) | 26 (38)
Vaginal odor (Pregnancy, puerperium and perinatal conditions) | 54 (84) | 25 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT02901626/Prot_SAP_ICF_000.pdf